CLINICAL TRIAL: NCT00711971
Title: Does EPA or DHA Prevent Depressive Symptoms in Pregnancy and Postpartum?
Brief Title: Does Fish Oil Prevent Depression in Pregnancy and Postpartum?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ellen Mozurkewich, Adjunct Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HUM00004684; R21AT004166-01A1 (NIH)
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EPA-rich fish oil supplement (Active Comparator): EPA-rich fish oil supplement
  Interventions: Drug: EPA-rich fish oil supplement
- DHA-rich fish oil supplement (Active Comparator): DHA-rich fish oil supplement
  Interventions: Drug: DHA-rich fish oil supplement
- Soy Oil placebo (Placebo Comparator): Soy oil
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: EPA-rich fish oil supplement — 1060 mg EPA plus 274 mg DHA
  Other Names: ProEPA Xtra
  Arms: EPA-rich fish oil supplement
Drug: DHA-rich fish oil supplement — 900 mg DHA plus 180 mg EPA
  Other Names: ProDHA
  Arms: DHA-rich fish oil supplement
Drug: placebo — control arm
  Arms: Soy Oil placebo

SUMMARY:
This study is designed to test whether an alternative medicine treatment, fish oil, will prevent depressive symptoms in pregnant and postpartum women who have been found to be at risk for depression. Epidemiologists have observed that people who live in countries where people on average eat a diet high in fish have a lower risk of depression than people who live in populations that eat less fish. Postpartum depression is also less common in these countries. The omega-3 fatty acids found in fish oil are thought to be responsible for this beneficial effect of eating fish. The two major omega-3 fatty acids found in fish are eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). DHA is an essential building block of the brain and nerve tissue. EPA may act to optimize the electrical signals between nerve cells and brain cells and may help the immune system to function well.

Some researchers have treated people who are already suffering from depression with fish oil. Some of these studies have shown a benefit for the fish oil treatment and others have not. These studies have tested EPA and DHA alone and in various combinations. Currently, it is not known whether EPA or DHA is more effective in preventing and treating depression. Some of the researchers involved in this study have learned how to identify mothers who are most at risk for developing depression during and after pregnancy. This study is designed to learn whether EPA-rich and DHA-rich fish oil supplements will prevent depressive symptoms in women who are at risk to develop depression.

ELIGIBILITY:
Inclusion Criteria:

* Women who are more than 12 weeks pregnant but less than 20 weeks pregnant
* Women who are found to be at risk for depression
* Women who have been treated for depression in the past
* Women with depression after a previous pregnancy
* Women planning to deliver at University of Michigan Hospital

Exclusion Criteria:

* Women who have major depression or other psychiatric disorders (current substance abuse, schizophrenia, bipolar disorder) at the time of screening
* Women who are currently taking anti-depressant or other psychiatric medications
* Women who routinely eat more than 2 fish meals per week
* Women on anticoagulants (blood thinners)
* Women currently taking omega-3 fatty acid dietary supplements (fish oil, flaxseed oil or cod liver oil)
* Women with bleeding disorders such as von Willebrand's disease
* Women under the age of 18
* Women with a multiple gestation (twins, for example)
* Women planning to deliver at another hospital
* Women planning to move away before 6 weeks after delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Mozurkewich, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Mozurkewich E, Chilimigras J, Klemens C, Keeton K, Allbaugh L, Hamilton S, Berman D, Vazquez D, Marcus S, Djuric Z, Vahratian A. The mothers, Omega-3 and mental health study. BMC Pregnancy Childbirth. 2011 Jun 22;11:46. doi: 10.1186/1471-2393-11-46. PMID 21696635
- [Result] Mozurkewich EL, Greenwood M, Clinton C, Berman D, Romero V, Djuric Z, Qualls C, Gronert K. Pathway Markers for Pro-resolving Lipid Mediators in Maternal and Umbilical Cord Blood: A Secondary Analysis of the Mothers, Omega-3, and Mental Health Study. Front Pharmacol. 2016 Sep 7;7:274. doi: 10.3389/fphar.2016.00274. eCollection 2016. PMID 27656142
- [Result] Williams JA, Romero VC, Clinton CM, Vazquez DM, Marcus SM, Chilimigras JL, Hamilton SE, Allbaugh LJ, Vahratian AM, Schrader RM, Mozurkewich EL. Vitamin D levels and perinatal depressive symptoms in women at risk: a secondary analysis of the mothers, omega-3, and mental health study. BMC Pregnancy Childbirth. 2016 Aug 3;16(1):203. doi: 10.1186/s12884-016-0988-7. PMID 27485050
- [Result] Romero VC, Somers EC, Stolberg V, Clinton C, Chensue S, Djuric Z, Berman DR, Treadwell MC, Vahratian AM, Mozurkewich E. Developmental programming for allergy: a secondary analysis of the Mothers, Omega-3, and Mental Health Study. Am J Obstet Gynecol. 2013 Apr;208(4):316.e1-6. doi: 10.1016/j.ajog.2013.01.024. PMID 23531329
- [Result] Mozurkewich EL, Clinton CM, Chilimigras JL, Hamilton SE, Allbaugh LJ, Berman DR, Marcus SM, Romero VC, Treadwell MC, Keeton KL, Vahratian AM, Schrader RM, Ren J, Djuric Z. The Mothers, Omega-3, and Mental Health Study: a double-blind, randomized controlled trial. Am J Obstet Gynecol. 2013 Apr;208(4):313.e1-9. doi: 10.1016/j.ajog.2013.01.038. PMID 23531328
- [Result] Ren J, Mozurkewich EL, Sen A, Vahratian AM, Ferreri TG, Morse AN, Djuric Z. Total Serum Fatty Acid Analysis by GC-MS: Assay Validation and Serum Sample Stability. Curr Pharm Anal. 2013;9(4):331-339. doi: 10.2174/1573412911309040002. PMID 25110470
- [Result] Berman D, Clinton C, Limb R, Somers EC, Romero V, Mozurkewich E. Prenatal Omega-3 Supplementation and Eczema Risk among Offspring at Age 36 Months. Insights Allergy Asthma Bronchitis. 2016;2(1):1. doi: 10.21767/2471-304X.100014. Epub 2016 Apr 10. PMID 28649675
- [Derived] England JA, Jain J, Holbrook BD, Schrader R, Qualls C, Mozurkewich E. Effect of prenatal EPA and DHA on maternal and cord blood insulin sensitivity: a secondary analysis of the mothers, omega 3, and mental health study. BMC Pregnancy Childbirth. 2019 Nov 29;19(1):452. doi: 10.1186/s12884-019-2599-6. PMID 31783739
- [Derived] Mozurkewich EL, Berman DR, Vahratian A, Clinton CM, Romero VC, Chilimigras JL, Vazquez D, Qualls C, Djuric Z. Effect of prenatal EPA and DHA on maternal and umbilical cord blood cytokines. BMC Pregnancy Childbirth. 2018 Jun 26;18(1):261. doi: 10.1186/s12884-018-1899-6. PMID 29940888

RESULTS

PARTICIPANT FLOW:
Groups:
- Soy Oil Placebo: Soy oil placebo: control arm
Period: Overall Study
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Started | 42 | 42 | 42
Completed | 39 | 38 | 41
Not Completed | 3 | 4 | 1
Not completed — Lost to Follow-up | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Population: All intent to treat - (all but lost to follow up) are included in baseline measures
Groups:
- Total: Total of all reporting groups
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo | Total
Number analyzed (Participants) | 39 | 38 | 41 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (5.0) | 30.6 (4.5) | 30.4 (5.9) | 30.3 (5.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 41 | 118
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33 | 29 | 34 | 96
  African-American | 4 | 4 | 2 | 10
  Hispanic-Latina | 0 | 4 | 3 | 7
  Asian | 1 | 1 | 1 | 3
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Native Hawaiian or other Pacific ethnicity | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 38 | 41 | 118
Gestational age at enrollment [Mean (Standard Deviation); unit: weeks] | 15.9 (2.6) | 17 (2.3) | 16.2 (2.3) | 16.36 (2.4)
Parity [Mean (Standard Deviation); unit: number of previous deliveries] | 0.87 (0.83) | 1.08 (0.94) | 0.85 (1.20) | 0.93 (1.01)
Past history of depression(self reported) [Number; unit: participants] | 32 | 30 | 33 | 95
BDI (Beck Depression Inventory) score [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory contains self-reported answers to questions concerning depression symptoms. It has been validated for use with pregnant women. Minimum score is 0 with 0 as no depression and maximum score is 63 representing the most severe depression.
  units on a scale | 8.41 (5.65) | 7.79 (5.29) | 7.15 (5.21) | 7.72 (5.38)
EPDS Screen (Edinburgh Prenatal Depression Scale) [Mean (Standard Deviation); unit: units on a scale] — The EPDS Screen is self-administered and subsequently scored by researchers on a 0 - 30 point range with 0 as no depression and 30 as most severe.
  units on a scale | 7.93 (4.63) | 7.56 (4.49) | 7.34 (4.40) | 7.80 (4.51)

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory
Description: The Beck Depression inventory scores depression based on 21 items, with a score of 0 - 3 on each item where 0 is no depression and a score of 31 or more is clinically depressed. The 21 items were summed to obtain the total score (The maximum possible score is 63.)
Time Frame: 6 - 8 weeks postpartum
Population: Per protocol analysis is reported here.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  BDI at 24-28 weeks' gestation | 7.9 (3.7) | 6.5 (4.7) | 6.3 (4.1)
  BDI at 34-36 weeks' gestation | 7.4 (5.0) | 5.9 (4.9) | 7.2 (5.2)
  BDI at 6-8 weeks postpartum | 6.6 (5.2) | 5.1 (4.4) | 6.2 (6.5)
Statistical Analysis 1: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Significance for the BDI test at 26-28 weeks; Test type: Superiority or Other; p = .29, ANOVA
Statistical Analysis 2: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Significance for BDI at 34-36 weeks gestation; Test type: Superiority or Other; p = .51, ANOVA
Statistical Analysis 3: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; BDI score at 6-8 weeks postpartum; Test type: Superiority or Other; p = .56, ANOVA

2. Other Pre Specified Outcome: Maternal Outcomes
Description: While the maternal outcomes assess criteria during pregnancy and relating to delivery they were assessed at visits 26 - 28 weeks gestational age, 34-36 weeks gestational age and at the post partum visit 6- 8 weeks after delivery.
Time Frame: visits at 26 - 28 weeks gestational age, 34-36 weeks gestational age during pregnancy and at the post partum visit 6- 8 weeks after delivery
Population: Gestational hypertension and diabetes were self-reported for all participants so her data is included for those two rows.
  One woman in the soy placebo arm delivered out of the geographic area, so documentation of delivery outcome is unavailable for analysis.
Measure: Number; unit: participants
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Number analyzed (Participants) | 39 | 38 | 41
participants
  Gestational Hypertension or Preeclampsia | 8 | 2 | 5
  Gestational Diabetes Mellitus | 7 | 1 | 2
  Induced Labor: number analyzed (Participants) | 39 | 38 | 40
  Induced Labor | 15 | 12 | 8
  Cesarean Section: number analyzed (Participants) | 39 | 38 | 40
  Cesarean Section | 10 | 12 | 11
  Spontaneous Vaginal Delivery: number analyzed (Participants) | 39 | 38 | 40
  Spontaneous Vaginal Delivery | 25 | 25 | 28
  Operative Vaginal Delivery: number analyzed (Participants) | 39 | 38 | 40
  Operative Vaginal Delivery | 4 | 1 | 1
Statistical Analysis 1: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Gestational diabetes mellitus; Test type: Superiority or Other; p = .06, Fisher Exact
Statistical Analysis 2: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Hypertension or preeclampsia; Test type: Superiority or Other; p = .12, Fisher Exact
Statistical Analysis 3: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Induced labor; Test type: Superiority or Other; p = .20, Fisher Exact
Statistical Analysis 4: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Cesarean section; Test type: Superiority or Other; p = .08, Fisher Exact
Statistical Analysis 5: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Spontaneous vaginal delivery; Test type: Superiority or Other; p = .88, Fisher Exact
Statistical Analysis 6: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Operative vaginal delivery; Test type: Superiority or Other; p = .32, Fisher Exact

3. Other Pre Specified Outcome: Gestational Age at Delivery (Weeks)
Time Frame: delivery date was assessed by medical record review between 1 day and 8 weeks after delivery
Population: Gestational age is measured based on the pregnancy not the neonates, therefore although there were 40 babies born to the 39 mothers randomized to the EPA-rich fish oil, it is proper to consider the participants analyzed to be the 39 participating mothers. This is clarified still further by identifying the units appropriately as pregnancies.
Measure: Mean (Standard Deviation); unit: weeks
Units Other Than Participants: pregnancies
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Number analyzed (Participants) | 39 | 38 | 41
Number analyzed (pregnancies) | 39 | 38 | 41
weeks | 39.1 (1.5) | 40.4 (0.9) | 39.1 (1.5)
Statistical Analysis 1: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Test type: Superiority or Other; p < .0001, ANOVA

4. Other Pre Specified Outcome: Estimated Blood Loss (ml)
Time Frame: Within 24 hours after delivery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Number analyzed (Participants) | 39 | 38 | 41
mL | 507 (481) | 508 (325) | 454 (296)
Statistical Analysis 1: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Test type: Superiority or Other; p = .81, ANOVA

5. Other Pre Specified Outcome: Neonatal Birthweight
Description: Mean weight in grams: where <2500 gm is considered small for gestational age and >4500 gm is considered large for gestational age.
Time Frame: immediately after birth
Population: Data is provided for all babies on whom delivery weights were available with a set of twins in EPA rich fish oil arm and a delivery elsewhere for whom no birth weight was available for one baby from a mother in the Soy oil placebo arm. Thus there is 1 more participant than mothers participating in the EPA-rich arm and one less in the soy oil arm.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Number analyzed (Participants) | 40 | 38 | 40
grams | 3402 (550) | 3774 (438) | 3309 (555)
Statistical Analysis 1: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Test type: Superiority or Other; p < .001, ANOVA; Kruskal-Wallis test was used for outliers; Tukey multiple comparisons test was also used

6. Other Pre Specified Outcome: NICU (Neonatal Intensive Care Unit) Admissions
Description: Admission to the NICU
Time Frame: 6 weeks post delivery
Population: One set of twins in group A
Measure: Count of Participants; unit: Participants
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Number analyzed (Participants) | 40 | 38 | 40
Participants | 6 | 2 | 4
Statistical Analysis 1: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Test type: Superiority or Other; p = .39, ANOVA

7. Other Pre Specified Outcome: One Minute Apgar Score
Description: Apgar scores are based on a scale of 0 - 10 where 0 is a dead baby and 10 is an optimally vigorous newborn. The Apgar score analyzed here is the one minute Apgar.
Time Frame: 1 minute after birth
Population: One set of twins from EPA group; Soy oil arm has data for only 40 as one baby was born elsewhere so Apgar data is not available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Number analyzed (Participants) | 40 | 38 | 40
units on a scale | 7.3 (2.2) | 7.9 (1.8) | 7.9 (1.9)
Statistical Analysis 1: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Test type: Superiority or Other; p = .19, ANOVA

8. Other Pre Specified Outcome: Five Minute Apgar Score
Description: Apgar scores are based on a scale of 0 - 10 where 0 is a dead baby and 10 is an optimally vigorous newborn. The Apgar score analyzed here is the five minute Apgar.
Time Frame: 5 minutes after birth
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Number analyzed (Participants) | 40 | 38 | 40
units on a scale | 8.6 (0.8) | 9.1 (0.2) | 8.9 (0.5)
Statistical Analysis 1: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Test type: Superiority or Other; p < 0.01, ANOVA

9. Other Pre Specified Outcome: Cord Arterial pH
Description: Arterial blood gas analysis of umbilical cord blood
Time Frame: Immediately after birth (collected within the first hour after delivery)
Population: Umbilical cord gases (pH) were sent at the discretion of the delivering physician and so were not available for all participants.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Number analyzed (Participants) | 34 | 31 | 31
pH | 7.26 (0.09) | 7.27 (0.05) | 7.27 (0.06)
Statistical Analysis 1: Comparison: EPA-rich Fish Oil Supplement vs DHA-rich Fish Oil Supplement vs Soy Oil Placebo; Test type: Superiority or Other; p = 0.54, ANOVA

ADVERSE EVENTS:
Time Frame: Up to 36 weeks (from enrollment at 12 - 20 weeks gestational age) through 6- 8 weeks after delivery
Description: The population listed as at risk here represents all 42 mothers randomized to each arm, but for NICU admissions and infant jaundice, the denominator (number at risk) represents the number of babies born to the mothers in each arm for whom data were available.
Arm/Group | EPA-rich Fish Oil Supplement | DHA-rich Fish Oil Supplement | Soy Oil Placebo
Serious Adverse Events (participants affected / at risk) | 8/42 | 5/42 | 5/42
Other Adverse Events (participants affected / at risk) | 28/42 | 23/42 | 22/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | EPA-rich Fish Oil Supplement (N=42) | DHA-rich Fish Oil Supplement (N=42) | Soy Oil Placebo (N=42)
Premature Delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
late miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Neonatal ICU Admission (Pregnancy, puerperium and perinatal conditions) | 6/40 (6) | 2/38 (2) | 4/41 (4)
Postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) | 0 (0)
Maternal ICU admission (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — Maternal ICU admission
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | EPA-rich Fish Oil Supplement (N=42) | DHA-rich Fish Oil Supplement (N=42) | Soy Oil Placebo (N=42)
Aftertaste (Gastrointestinal disorders) | 7 | 8 | 7 — Aftertaste (sometimes described as fishy, as lemon, as strawberry or just "aftertaste"
Belching (Gastrointestinal disorders) | 11 | 14 | 12
Gestational Diabetes (Endocrine disorders) | 5 | 0 | 1
Infant Jaundice (Blood and lymphatic system disorders) | 9/40 | 3/38 | 2/41
Loose stools (Gastrointestinal disorders) | 5 | 2 | 5
mastitis (Reproductive system and breast disorders) | 0 | 4 | 0
nausea (Gastrointestinal disorders) | 4 | 1 | 2
Preterm Contractions (Reproductive system and breast disorders) | 4 | 4 | 1
Heartburn (Gastrointestinal disorders) | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes